CLINICAL TRIAL: NCT02386332
Title: A Randomized Multicenter Study Comparing Unrelated Umbilical-cord Blood Transplant Versus Human Leukocyte Antigen (HLA)-Haploidentical Related Hematopoietic Stem Cell Transplant for Adult Patients With Hematologic Malignancies
Brief Title: A Randomized Multicenter Study to Compare Two Types of Transplant in Adult Patients With Hematologic Malignancies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Other Study IDs: TPH
Record Dates: First submitted 2015-02-26; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Transplantation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- umbilical cord blood transplant (UCBT): Patients to receive umbilical cord blood transplant (UCBT) are conditioned with the myeloablative conditioning regimen (preparative therapy with thiotepa, fludarabine, intravenous busulfan and anti-thymocyte globulin.). Also receive GVHD prophylaxis with cyclosporine A and prednisone and Additional Supportive Care
  Interventions: Procedure: transplantation
- HLA-haploidentical hematopoietic stem cell transplantation: Patients to receive HLA-haploidentical hematopoietic stem cell transplantation are conditioned with the myeloablative conditioning regimen (preparative therapy with thiotepa, fludarabine, intravenous busulfan). Also receive GVHD prophylaxis with cyclophosphamide, cyclosporine A and mycophenolate mofetil and Additional Supportive Care
  Interventions: Procedure: transplantation

INTERVENTIONS:
Procedure: transplantation

SUMMARY:
This is an open-label, prospective, observational, multicenter, randomized study to compare the efficacy between unrelated umbilical cord blood transplantation (UCBT) and HLA-haploidentical related hematopoietic stem cell transplantation ,after myeloablative conditioning for adult patients with hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Age: subjects ≥ 18 and ≤ 55 years old.
2. Patients without suitable matched related donor
3. Diagnosed with acute leukemia or myelodysplastic syndrome in which allogeneic transplantation is considered the most potentially curative therapeutic option.
4. Written consent form signed.

Exclusion Criteria:

* Performance status: Eastern Cooperative Oncology Group(ECOG) score >2
* Prior allogenic hematopoietic stem cell transplant
* Left-ventricular ejection fraction at rest < 45%, uncontrolled arrhythmias or symptomatic heart failure.
* Diffusing capacity (DLCO) and/or forced vital capacity (FVC) < 39% of predicted values or symptomatic pulmonary disease
* Altered liver function tests (total bilirubin > 2 mg/dL and/or alanine aminotransferase, aspartate aminotransferase , and or active hepatitis or cirrhosis.
* Serum creatinine > 2 mg/dL or estimated creatinine clearance < 50 mL/min
* Evidence of uncontrolled bacterial, viral or fungal infection prior to the conditioning regimen
* Serious diseases that prevent patients from receiving chemotherapy treatments.
* Concomitant neoplasms.
* Pregnancy or breast-feeding.
* Any other medical, surgical or psychiatric condition that is considered by the attending and/or medical team as a contraindication for intensive treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Diagnosed with acute leukemia or myelodysplastic syndrome in which allogeneic transplantation is considered the most potentially curative therapeutic option
Sampling Method: Probability Sample
Enrollment: 206 (Estimated)
Dates: Start 2015-03; Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Sanz, MD, Study Chair — University Hospital La Fe, Valencia